CLINICAL TRIAL: NCT07356297
Title: Comparing Remotely-delivered Interventions to Promote Cessation Among Adults Who Smoke Menthol Cigarettes
Brief Title: Remote Interventions for Menthol Cigarette Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lara Coughlin, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00275412; SU-2024C2-40036 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quitline (QL) (Active Comparator): Participants complete QL services
  Interventions: Behavioral: Quitline (QL)
- Quitline (QL) + App (Active Comparator): Participants complete QL services and download our incentive-based mobile app
  Interventions: Behavioral: Quitline (QL); Behavioral: Mobile incentive-based intervention

INTERVENTIONS:
Behavioral: Quitline (QL) — QL services include scheduled and on-demand phone and digital interactions with a coach, as well as optional ancillary services and nicotine replacement therapy by mail.
Behavioral: Mobile incentive-based intervention — The app-based intervention incentivizes participants for daily check-ins, smoking cessation, and QL calls. Participants also receive encouragement to set a smoking quit date from a study interventionist and receive motivational messages in the app.
  Arms: Quitline (QL) + App

SUMMARY:
The purpose of this study is to evaluate whether a digital, incentive-based program, used in conjunction with traditional quitline (QL) services, can be beneficial to quitline callers who smoke menthol cigarettes. The services evaluated focus on coaching, support, and/or incentives for individuals who wish to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* adults (ages 18+) who call partnered quitlines (QL); and
* currently smoke menthol cigarettes; and
* are fluent in English; and
* plan to live in the United States for the full trial duration; and
* have daily smartphone access (including data access) or are willing to use a study-provided smartphone and data plan
* ability to provide informed consent

Exclusion Criteria:

* not ready to set a quit date within 30 days; or
* have not smoked in the past 7 days
* Inability to speak/understand English
* Conditions precluding informed consent or understanding of intervention or assessment content
* PI discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | 3-, 6-, 9- and 12- months post baseline
  Participants will self-report (yes/no) past 30-day combustible tobacco use.

SECONDARY OUTCOMES:
Smoking Cessation With Lapses | 3-, 6-, 9- and 12- months post baseline
  Participants will self-report of cessation from combustible tobacco products, with the exception of up to 5 cigarettes (lapses), since 2 weeks after their quit date (i.e., 2 week "grace period").

CONTACTS AND LOCATIONS:
Overall Officials: Lara Coughlin, PhD, Principal Investigator — University of Michigan; Erin Bonar, PhD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: Yes
Consistent with sponsor requirements, de-identified data will be shared with the Patient Centered Outcomes Research Institute (PCORI), its collaborators, and associated research partners.
Supporting Information: Study Protocol, SAP, ICF